CLINICAL TRIAL: NCT01450046
Title: A Phase I Dose-Escalation Study of the Safety and Pharmacokinetics of Vitamin E δ-Tocotrienol Following Multiple Dose Administration in Healthy Subjects
Brief Title: Vitamin E δ-Tocotrienol Multiple Dose in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); BioGene Life Science (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MCC-16153
Record Dates: First submitted 2011-10-07; First posted 2011-10-12 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-07

CONDITIONS: Pancreatic Cancer
Keywords: pancreas; gastrointestinal; GI; prevention; vitamin E
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — tocotrienol, delta

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Phase I Dose Escalation (Experimental): Each investigator will be provided with adequate supplies of Vitamin E δ -Tocotrienol, which will be supplied as 100-mg, 200-mg, and 400-mg capsules. Vitamin E δ-Tocotrienol will be administered orally once. The dose administered to each subject will be fixed and based on cohort assignment. Doses will be administered at the clinical site during each protocol-defined visit.
  Interventions: Drug: Vitamin E δ-Tocotrienol

INTERVENTIONS:
Drug: Vitamin E δ-Tocotrienol — Vitamin E δ-Tocotrienol will be administered orally as a single agent twice daily for 14 consecutive days. Vitamin E δ-Tocotrienol is supplied as 100-mg, 200-mg, and 400-mg capsules. The first cohort will be dosed with δ-tocotrienol at 100 mg twice daily for 14 consecutive days. A minimum of 3 subjects is planned for each dosing cohort with Vitamin E δ-Tocotrienol dose escalation dependent on safety and available PK data from prior cohorts. At the MTD or MAD, 18 subjects will be enrolled.
  Other Names: Delta-tocotrienol

SUMMARY:
The Principal Investigator believes that Vitamin E δ-Tocotrienol will slow the progression of pancreatic cancer cells. Therefore, the investigators must determine the safety and tolerability of Vitamin E δ-Tocotrienol in healthy participants before administering to cancer patients. The investigators will do this by giving participants a dose of up to1600 mg twice a day, not to exceed 3200 mg total for 14 consecutive days.

DETAILED DESCRIPTION:
Participants will be accrued in cohorts of three. The decision to dose escalate will be made by the Cohort Review Committee (CRC) based on safety after the last subject in the current cohort has completed the Study Treatment Period. The study will consist of the following procedures:

* Pre-Treatment Period: The screening period must occur within 7 days of dosing.
* Study Treatment Period (14 days): Vitamin E δ-Tocotrienol will be administered orally twice daily for 14 consecutive days
* Post-Treatment Period: Subject will return to the study site 7 days after the dose of Vitamin E δ-Tocotrienol for an end-of-treatment assessment. On day 8 (± 2 days) after the last dose of study drug, the investigator will obtain follow-up information. Any serious adverse events (SAEs) present at 7 days after the last dose and possibly related to study drug will be followed until resolution, stabilization, or initiation of treatment that confounds the ability to assess the event.

ELIGIBILITY:
Inclusion Criteria:

* Equal to or greater than 18 years of age
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤2
* Adequate organ function:

  * Serum creatinine ≤1.5 mg/dL or calculated creatinine clearance ≥60 mL/min.
  * Bilirubin ≤ the intuitional upper limits of normal
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) to be within institutional normal range
  * Absolute neutrophil count (ANC) ≥1000mm³
  * Platelet count ≥100,000mm³
* Has the capability of understanding the informed consent document and has signed the informed consent document
* Sexually active participants (male and female) must use medically acceptable methods of contraception during the course of the study.
* Women of childbearing potential must have a negative pregnancy test at screening.
* Able to understand and comply with the requirements of the protocol

Exclusion Criteria:

* receiving investigational therapy (other than the investigational therapy under study)
* Have received investigational therapy within 30 days prior to first dose of study drug
* Patients who are unable to swallow capsules
* Patients with prior malignancies, other than squamous or basal cell carcinomas, unless disease free for ≥ 5 years
* Have had prior major surgery within 30 days prior to first dose of study drug
* The patient has active infection or fever >38.5C within 3 days prior to first dose of study drug.
* Have uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, hypertension, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Unable or unwilling to stop taking vitamins, herbal remedies, or nonprescription medications
* Pregnant or breastfeeding
* Unable or unwilling to abide by the study protocol or cooperate fully with the investigator or designee

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-10; Primary Completion 2013-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment Related Adverse Events | 3 Weeks Per Participant
  The primary objective of this study is to evaluate the safety and tolerability of Vitamin E δ-Tocotrienol and to determine the maximum administered dose (MAD) or maximum tolerated dose (MTD) of Vitamin E δ-Tocotrienol administered twice daily for 14 days. Safety analyses and summary tables will include data collected for all subjects who receive at least one dose of study drug.

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of Vitamin E δ-Tocotrienol | 3 Weeks Per Participant
  To determine the effects of dose on the plasma pharmacokinetic (PK) of Vitamin E δ-Tocotrienol following multiple dose administration in healthy subjects.
Pharmacodynamic (PD) Markers of Vitamin E δ-Tocotrienol Activity in Peripheral Blood | Day 1, Day 8 Day 14
  Peripheral blood mononuclear cells will be collected at each time point for examination of biomolecular markers not limited to Erk, p-Erk, AKT, p-AKT, p27, Ki-67, and exportin.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Klapman, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States